CLINICAL TRIAL: NCT04437173
Title: Immersive Audiovisual Distraction With Virtual Reality (VR) to Reduce Anxiety and Sedation Requirements During Pain Procedures in the Interventional Pain Clinic
Brief Title: Pain Procedures and Anxiolysis Via Distraction With Virtual Reality
Acronym: PAIN-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1480456
Record Dates: First submitted 2020-06-09; First posted 2020-06-18 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Virtual Reality; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Arm (Experimental): Patients undergo interventional pain procedure with virtual reality distraction
  Interventions: Device: Virtual Reality Headset Distraction
- No Intervention Arm (No Intervention): Patients undergo interventional pain procedure without virtual reality distraction

INTERVENTIONS:
Device: Virtual Reality Headset Distraction — Patient wears a virtual reality headset during interventional pain procedure
  Arms: Virtual Reality Arm

SUMMARY:
The purpose of this study is to evaluate the efficacy of VR distraction on reducing anxiety patients undergoing interventional pain procedures compared to placebo/active placebo or a non VR option.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years old, who are referred to University of California Davis Pain Medicine Clinic and require an interventional pain procedure
* English speaking
* Having the ability to understand oral and written instructions
* Willing to fill out psychometric surveys.

Exclusion Criteria:

* Pregnant women
* Prisoners
* Patients who have high risk of motion sickness, seizure disorder, or visual/hearing impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Anxiety Score | Immediately before procedure and immediately after procedure.
  State-Trait Anxiety Inventory (Self-reported anxiety instrument containing two separate 2-item subscales that measure trait (baseline) and state (situational) anxiety; Total range 20 to 80 with higher scores indicating greater anxiety)

SECONDARY OUTCOMES:
Pain Score | Immediately before procedure, during procedure, and immediately after procedure
  Pain score on an 11-point numerical rating scale (Total range 0-10 with higher scores indicating greater pain)
Sedation Requirements | During course of procedure
  Amount of benzodiazepines and opioid medications given
Global Impression of Change | Immediately after procedure
  Global Impression of Change on a 7-point scale (Lower scores indicating decline in clinical status, and higher scores indicating improvement in clinical status)
Patient Experience Satisfaction | Immediately after procedure
  Experience Satisfaction on an 11-point scale (Total range 0-10 with higher scores indicating higher patient experience satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Naileshni Singh, MD, Principal Investigator — University of California, Davis; John Sun, MD, Principal Investigator — University of California, Davis; Michael Jung, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Interventional Pain Clinic, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No